CLINICAL TRIAL: NCT04422249
Title: A RCT Study of Laparoscopic Middle Hepatic Vein Guidance and Traditional Anatomic Hemihepatectomy
Brief Title: A Study of Laparoscopic Middle Hepatic Vein Guidance and Traditional Anatomic Hemihepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SWHZSG009
Record Dates: First submitted 2020-05-20; First posted 2020-06-09 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Laparoscopic Middle hepatic vein Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Two different treatments are conducted on the participant base on the randomized choices
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic middle hepatic vein guidance hemihepatectomy (Experimental): In theory, the advantages of anatomical hemihepatectomy guided by middle hepatic vein are as follows: 1) correctly guiding the transecting plane of the liver parenchyma can reduce the cross-sectional area of the liver and avoid damaging the vascular ducts of the pre-cut liver. so as to reduce the residue of necrotic tissue without blood supply and reduce the occurrence of postoperative complications. 2) active anatomy and exposure of hepatic vein can avoid uncontrollable bleeding after passive injury of hepatic vein, and laparoscopic anatomy has obvious advantage in exposing hepatic vein. 3) it may reduce the early recurrence rate of hepatocellular carcinoma after operation.
  Interventions: Procedure: laparoscopic middle hepatic vein guidance anatomic hemihepatectomy
- laparoscopic traditional anatomic hemihepatectomy (Active Comparator): According to textbooks and the views of some scholars at present, traditional anatomical hepatectomy (non-hepatic vein-guided anatomical hepatectomy) has the following advantages: 1) avoiding exposure of hepatic vein can reduce the probability of injury to the trunk of hepatic vein, thus reduce the risk of massive bleeding during operation; 2) the difficulty of operation is relatively low, and a better short-term and long-term effect can be obtained.
  Interventions: Procedure: laparoscopic middle hepatic vein guidance anatomic hemihepatectomy

INTERVENTIONS:
Procedure: laparoscopic middle hepatic vein guidance anatomic hemihepatectomy — 95 patients with primary HCC were divided into the middle hepatic vein guidance group(n=45) and the traditional group(n=45) according to the odd and even Numbers, and sealed into envelopes.Outcomes were monitored and evaluated during the 3-year follow-up period
  Other Names: laparoscopic traditional anatomic hemihepatectomy

SUMMARY:
The study, entitled "RCT study of laparoscopic middle hepatic venous guidance versus conventional ananatomical hemihepatectomy", was designed to compare the efficacy of two different ananatomical hemihepatectomy procedures under laparoscopy.

DETAILED DESCRIPTION:
Backgroud & Aim:Hepatectomy is the main way to treat all kinds of liver surgical diseases, which can be divided into anatomic hepatectomy and non-anatomic hepatectomy.Among them, anatomic hepatectomy is suitable for primary liver cancer, hepatolithiasis and other benign and malignant diseases;It can be divided into hepatic venous guidance and non-hepatic venous guidance hepatectomy (traditional ananatomical hepatectomy).The aim of this study was to observe and compare the perioperative period and follow-up results of the two different laparoscopic surgical resection methods, and to provide high-level evidence-based medicine evidence for the selection of surgical methods for laparoscopic anatomical hemihepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. the site was limited to the patients who were suitable for dissecting hemihepatectomy；
2. the type of disease was limited to hepatocellular carcinoma；
3. the patients were generally able to tolerate anesthesia, the liver reserve function was good, and the patients were suitable for laparoscopic surgery；
4. child-pugh grade A, no severe liver cirrhosis, portal hypertension, no extrahepatic and extrahepatic metastasis and main vascular invasion；
5. the subjects who participated in this study indicated that they were willing to accept the two surgical methods and agreed to be randomly divided into groups during the operation；
6. 18 ≤ age ≤ 70, male or female.

Exclusion Criteria:

1. preoperative liver function Child-pugh grade B or C;
2. patients with poor general condition and could not tolerate pneumoperitoneum or anesthesia;
3. patients with severe liver cirrhosis, portal hypertension and lesions invading liver porta;
4. patients with other treatment methods such as radio frequency ablation in addition to dissecting hepatectomy;
5. repeated abdominal operations resulting in severe abdominal adhesion, unable to perform laparoscopic hepatectomy; male and female are not limited

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 3 years
  follow-up after the surgery every 3 months, to understand statistics 1-year overall survival、3-year overall survival、1-year disease-free survival、3-year disease-free survival

SECONDARY OUTCOMES:
Perioperative results | Duration perioperation(an expected average of 3 days)
  the angle of hepatic vein between segment Ⅳ b and Ⅴ, angle between MHV and IVC
intraoperative parameters | during the operation
  blood loss per unit area will be combined to report intraoperative parameters in milliliter/square centimetre(ml/c㎡）

OTHER OUTCOMES:
Incidence of postoperative complications | Duration hospitalization(an expected average of 7 days)
  hemorrhage,biliary leakage,ascites,intra-abdominal infection,pleural effusion,pulmonary infection,cardiopulmonary insufficiency，liver function failure

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China